CLINICAL TRIAL: NCT05023746
Title: Clinical Evaluation of Genetron Lung Cancer Panel in Non-small Cell Lung Cancer Patients
Status: Completed | Type: Observational
Sponsor: Genetron Health (Industry)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); The Second Affiliated Hospital Zhejiang University School of Medcine (Unknown); Henan Cancer Hospital (Other Government); The First Hospital of Jilin University (Other); Genetron Health (Beijing) Co., Ltd. (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2019071915080046
Record Dates: First submitted 2021-08-11; First posted 2021-08-27 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Clinically diagnosed as non-small cell lung cancer samples
  Interventions: Diagnostic Test: Genetron lung cancer panel

INTERVENTIONS:
Diagnostic Test: Genetron lung cancer panel — Follows the principle of synchronous blinding. The enrolled cases are coded, and the enrolled samples are detected with Genetron lung cancer panel and comparison methods. The detection results are compared, and the samples that are inconsistent with the detection results of similar products on the market are reviewed by the the Sanger sequencing method, when the site detection results compared with Sanger sequencing method are inconsistent, Sanger's detection results are recognized. The results were determined independently according to the cutoff values or interpretation requirements provided by each method, and relevant statistics were used to evaluate clinical application performance of Genetron lung cancer panel.

SUMMARY:
The purpose of this trail is to evaluate the performance of Genetron lung cancer panel in non-small cell lung cancer patients using semiconductor sequencing method.

DETAILED DESCRIPTION:
This trial follows the principle of synchronous blinding. The enrolled cases are coded, and the enrolled samples are detected with Genetron lung cancer panel and comparison methods. The detection results are compared, and the samples that are inconsistent with the detection results of similar products on the market are reviewed by the the Sanger sequencing method, when the site detection results compared with Sanger sequencing method are inconsistent, Sanger's detection results are recognized. The safety and effectiveness of this panel are confirmed and evaluated. Meanwhile, the accuracy of this panel for the following drug companion diagnostic tests: EGFR gene 19 exon deletion and L858R point mutation in gefitinib tablets, erlotinib hydrochloride and icotinib hydrochloride tablets, T790M point mutation in methanesulfonate acid osimertinib tablets, ALK gene fusion in crizotinib capsules.

The results were determined independently according to the cutoff values or interpretation requirements provided by each method, and relevant statistics were used to evaluate clinical application performance of Genetron lung cancer panel.

ELIGIBILITY:
Inclusion Criteria:

1. Cancer samClinically diagnosed as non-small cell lung samples (mainly lung adenocarcinoma and some lung squamous cell carcinoma, adenosquamous carcinoma, large cell carcinoma, etc.), and a small number of other cancer types are enrolled as interference samples.
2. Collect some samples of relevant medical information before and after the use of targeted drugs. This part of the samples should have relevant previous molecular diagnosis results.
3. Able to provide samples in time according to the requirements of the plan: samples for DNA/RNA extraction: 10 pieces of 10 µm thickness for each sample or 10 pieces of paraffin rolls. Samples for FISH experiment: 5 slices of 3-4µm thickness.
4. The pathological examination conforms to the types of tissue samples listed in the above table. The HE staining results show that the tumor content is not less than 50%, and the paraffin slice damage should be avoided.
5. The sample should have corresponding basic clinical information, including: patient visiting number/medical record number/specimen number, age, gender, pathological diagnosis result, molecular diagnosis result (if any).

Exclusion Criteria:

* Those who do not meet any of the above conditions are excluded. Reason: The included non-small cell lung adenocarcinoma samples and normal samples should have statistical significance, and the conclusions obtained should be scientific and valid. The selection of subjects for this study, while excluding research-related influencing factors, has no adverse effect on the health of the subjects.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospital sample
Sampling Method: Non-Probability Sample
Enrollment: 1052 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2019-09-17 (Actual)

PRIMARY OUTCOMES:
Efficacy of Genetron Lung Cancer Panel | 2 months
  The main purpose of this study is: by evaluating the Genetron Lung Cancer Panel to compare the results of simultaneous detection with similar products on the market and the Sanger sequencing method, and to calculate the coincidence rate and consistency of the panel and the comparison method.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - The First Hospital of Jilin University, Jilin
  - The Second Affiliated Hospital Zhejiang University School of Medcine, Zhejiang
  - Henan Cancer Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-07): https://cdn.clinicaltrials.gov/large-docs/46/NCT05023746/Prot_SAP_000.pdf